CLINICAL TRIAL: NCT06114524
Title: Effect of Binaural Beats on Level of Anxiety and Toleration in Patients Undergoing Upper Gastrointestinal Endoscopy Without Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, selim demirci, medical doctor, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Binaural
Record Dates: First submitted 2023-10-25; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Patient Satisfaction; Anxiety State; Tolerance
MeSH Terms: conditions — Patient Satisfaction; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- binaural music group (Experimental): Binaural music therapy was applied for 15 min before the procedure.
  Interventions: Other: binaural music
- control (No Intervention): The control group was kept in a quiet room for 15 minutes before the procedure and then taken for the procedure.

INTERVENTIONS:
Other: binaural music — In the binaural music group, an MP3 player and in-ear stereo headphones were provided. Music therapy was applied for 15 min before the procedure.
  Arms: binaural music group

SUMMARY:
To investigate the anxiolytic effects of binaural beat-embedded audio in patients undergoing sedation-free upper gastrointestinal endoscopy

DETAILED DESCRIPTION:
The study was conducted with the participation of 96 patients who were referred for endoscopy for various reasons. Data were collected by two researchers. Patients between the ages of 18-70 who had scheduled upper gastrointestinal endoscopy appointments were included in the study, regardless of gender and underlying diseases. Patients who had undergone endoscopic procedures before, were using medication for anxiety and panic disorders, required urgent endoscopic intervention, had advanced dementia, had hearing problems, had anatomical or inflammatory disorders in the external ear canals, and those who did not want to listen to music for 15 minutes before the procedure were not included in the study.

ELIGIBILITY:
Inclusion Criteria:

- Between 18-70 years old who had scheduled upper gastrointestinal endoscopy appointments

Exclusion Criteria:

* Anxiety and panic disorders
* Urgent endoscopic intervention
* Advanced dementia
* Hearing problems
* Anatomical or inflammatory disorders in the external ear canals

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | Within 20 minutes pre-procedure and 5 minutes after the procedure
  Comparative results of the differences in STAI scores before and 5 minutes after the endoscopy in the music and control groups. The State-Trait Anxiety Inventory (STAI) is a valid, self-report measure that consists of 40 items, with 20 items assessing state anxiety (STAI-S) and the other 20 items assessing trait anxiety (STAI-T). For both state and trait components, scores range from 20 to 80, with higher scores indicating higher levels of anxiety

SECONDARY OUTCOMES:
Patient satisfaction | 5 minutes after the procedure
  After the procedure, the patients were asked a series of questions for procedure evaluation (worse than expected, as expected, better than expected) and their willingness to have endoscopy again for their health (no, yes). The binaural music group was asked a three-item question with "yes-not sure-no" responses, inquiring whether the music increased relaxation and if they would like to listen to the same music again during a repeat procedure.
Heart rate | Within 20 minutes pre-procedure and 5 minutes after the procedure
  The comparison of heart rate in the music and control groups
Blood pressure | Within 20 minutes pre-procedure and 5 minutes after the procedure
  The comparison of systolic and diastolic blood pressure in the music and control groups
patient tolerance | During the procedure
  The patient's tolerance during the procedure was assessed by the physician using a scale as follows: 0 (complete tolerance during the procedure, only retching during endoscope insertion); 1 (retching less than 2 times during the procedure); 3 (retching 3 or more times during the procedure); 4 (attempt to remove the endoscope during the procedure).

CONTACTS AND LOCATIONS:
Locations (1):
- Abdurrahman Yurtaslan Oncology and Training Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Opartpunyasarn P, Vichitvejpaisal P, Oer-Areemitr N. The effect of binaural beat audio on anxiety in patients undergoing fiberoptic bronchoscopy: A prospective randomized controlled trial. Medicine (Baltimore). 2022 Jun 17;101(24):e29392. doi: 10.1097/MD.0000000000029392. PMID 35713444
- [Result] Isik BK, Esen A, Buyukerkmen B, Kilinc A, Menziletoglu D. Effectiveness of binaural beats in reducing preoperative dental anxiety. Br J Oral Maxillofac Surg. 2017 Jul;55(6):571-574. doi: 10.1016/j.bjoms.2017.02.014. Epub 2017 Mar 18. PMID 28325532
- [Result] Padmanabhan R, Hildreth AJ, Laws D. A prospective, randomised, controlled study examining binaural beat audio and pre-operative anxiety in patients undergoing general anaesthesia for day case surgery. Anaesthesia. 2005 Sep;60(9):874-7. doi: 10.1111/j.1365-2044.2005.04287.x. PMID 16115248
- [Derived] Demirci S, Sezer S. Effect of Binaural Beats on Anxiety and Tolerance in Patients Undergoing Upper Gastrointestinal Endoscopy Without Sedation: A Randomized Controlled Trial. J Integr Complement Med. 2024 Dec;30(12):1209-1216. doi: 10.1089/jicm.2023.0804. Epub 2024 Aug 1. PMID 39088370